CLINICAL TRIAL: NCT03719586
Title: A Multicenter, Multi-Outbreak, Randomized, Controlled Safety and Efficacy Study of Investigational Therapeutics for the Treatment of Patients With Ebola Virus Disease
Brief Title: Investigational Therapeutics for the Treatment of People With Ebola Virus Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 190003; 19-I-0003
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-11

CONDITIONS: Ebola Virus
Keywords: EBOV; Viral Hemorrhagic Fever; Ebola Treatment Center; Filovirus; Zaire Ebola Virus
MeSH Terms: conditions — Hemorrhagic Fevers, Viral | interventions — ZMapp; remdesivir; ansuvimab; atoltivimab, maftivimab, and odesivimab-ebgn drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A (Experimental): Remdesivir plus optimized Standard of Care (oSOC)
  Interventions: Drug: Remdesivir
- B (Experimental): MAb114 plus optimized Standard of Care (oSOC)
  Interventions: Drug: MAb114
- C (Experimental): REGN-EB3 plus optimized Standard of Care (oSOC)
  Interventions: Drug: REGN-EB3
- Control (Experimental): Zmapp plus optimized Standard of Care (oSOC)
  Interventions: Drug: ZMapp

INTERVENTIONS:
Drug: ZMapp — Three doses of 50 mg/kg of body weight administered intravenously every third day beginning on Day 1
  Arms: Control
Drug: Remdesivir — Administered intravenously with a loading dose on Day 1 (200 mg for adults and pediatric patients with body weight >= 40 kg and for pediatric patients weighing < 40 kg one loading dose of remdesivir 5 mg/kg) followed by 9 to 13 days of once-daily maintenance dosing starting on Day 2 and extending through Day 10 to 14 (100 mg for adults and pediatric patients with body weight >= 40 kg and for pediatric patients weighing < 40 kg remdesivir 2.5 mg/kg)
  Arms: A
Drug: MAb114 — 50 mg/kg of body weight administered intravenously on Day 1 as a single infusion
  Arms: B
Drug: REGN-EB3 — 150 mg/kg of body weight administered intravenously on Day 1 as a single infusion
  Arms: C

SUMMARY:
Background:

Ebola virus can cause serious illness or death. No medicines are approved to treat it. Researchers need to test new medicines to see if they help people recover from Ebola and are safe to give. They need to test the drugs and compare them in a controlled way. Researchers want to test 4 drugs with people who have Ebola and are in treatment centers.

Objective:

To study the safety and effectiveness of 4 drugs for people with Ebola virus.

Eligibility:

People of any age with Ebola infection who are in treatment centers

Design:

Participants will be screened with questions, medical history, and blood tests.

Participants will be randomly assigned to get 1 of 3 study drugs:

* ZMapp by IV over about 4 hours. It will be given 3 times, 3 days apart.
* Remdesivir by IV over about 1 hour. It will be given once a day for 10 days.
* Mab114 by IV for 30-60 minutes. It will be given 1 time.
* REGN-EB3 by IV for about 2 hours. It will be given 1 time.

For at least a week, participants will stay in isolation in a clinic. They will:

* Get supportive care and be monitored
* Have a small plastic tube (IV) put in an arm vein for several days to give fluids and collect blood.
* Get their study drug.
* Be monitored for disease signs and drug side effects. They may get medicines for side effects.
* Have blood and urine tests.

Participants will stay in the clinic until they finish the study drug and are well enough to leave.

Participants will have 2 follow-up visits over 2 months. They will answer questions and give blood and semen samples.

...

DETAILED DESCRIPTION:
Species Zaire ebolaviruses (EBOV) are members of the Filoviridae and are known primarily as the underlying cause of severe viral hemorrhagic fevers with disturbingly high case fatality rates. Between 1994 and the present, there have been many filovirus outbreaks affecting mostly central Africa, with 2 large outbreaks in 1995 in Kikwit, Democratic Republic of Congo (DRC), and in Gulu, Uganda in 2000-2001. The 2013-2016 West African outbreak significantly exceeded all previous outbreaks in geographic range, number of patients affected, and in disruption of typical activities of civil society. In 2018 there have been two additional outbreaks of EBOV infection, both in the Democratic Republic of the Congo and constituting the 9th and 10th recorded outbreaks of this infection in that country. The 10th outbreak is currently ongoing in the DRC as of December 2018 and has raised great concern because of the potential to expand greatly in scope and to spread to surrounding regions.

It has been suggested that one of the most important elements necessary to improve survival from Ebola virus infection is the provision of supportive care inclusive of hemodynamic support in the form of aggressive fluid replacement, ability to diagnose and correct severe metabolic derangements, early treatment of sepsis, and other standards of modern medical care. A small number of investigational therapeutics have been developed as putative antiviral strategies for treating this infection. Unfortunately, phase 1/2 data supporting the safety and efficacy of these agents are often limited, and thus there remains some degree of equipoise as to which of these interventions should be prioritized in the treatment of severe infection. The triple monoclonal antibody product ZMapp was studied through a randomized controlled trial (RCT) in the 2014-2016 West African outbreak and remains perhaps the best characterized of the available investigational products, but the end of that outbreak forced the RCT to close prior to crossing pre-specified evidentiary boundaries.

A WHO Research and Development Ebola Therapeutics Committee has agreed that, given the lethality of Ebola virus and the combination of human and non-human primate (NHP) efficacy data for ZMapp, either ZMapp+oSOC or oSOC alone could potentially be positioned as the control arm in comparative trials depending upon the preferences of the host countries. The DRC has chosen to use ZMapp + oSOC in the current protocol. However, both the nature and number of control and invegstigational arms may change over the course of the trial. Such changes would require protocol amendments.

This multicenter, multi-outbreak, randomized controlled trial will study the comparative safety and efficacy of additional investigational therapeutics compared to ZMapp in patients with known EBOV disease (Zaire) receiving oSOC. The primary endpoint of this comparison will be mortality by Day 28, with a number of secondary endpoints also planned that should generate important knowledge about the safety, ease of administration, and antiviral activity of all of these investigational interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males or females of any age with documented positive RT-PCR in blood for acute Ebola virus infection within 3 days prior to enrollment and who have symptoms of any duration.
* Willingness of study participant to accept randomization to any assigned treatment arm.
* All males and females of childbearing potential must be willing to use effective methods of contraception, from time of enrollment until Day 58 of study.
* Must agree not to enroll in another study of an investigational agent prior to completion of Day 28 of study.
* Ability to provide informed consent personally, or by a legally acceptable representative if the patient is unable to do so.

EXCLUSION CRITIERA:

* Patients who, in the judgment of the investigator, will be unlikely or unable to comply with the requirements of this protocol through Day 28.
* Prior treatment with any investigational antiviral drug therapy against Ebola virus infection within 5 half-lives or 30 days, whichever is longer, prior to enrollment. (Patients who have received an experimental (or, in future, potentially a licensed) immunization against Ebola virus remain eligible.)

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Ebola Treatment Centers throughout the DRC, Kinshasa Gombe, Democratic Republic of the Congo

REFERENCES:
- [Derived] Ottoni MP, Ricciardone JD, Nadimpalli A, Singh S, Katsomya AM, Pokoso LM, Petrucci R. Ebola-negative neonates born to Ebola-infected mothers after monoclonal antibody therapy: a case series. Lancet Child Adolesc Health. 2020 Dec;4(12):884-888. doi: 10.1016/S2352-4642(20)30278-9. PMID 33217357
- [Derived] Mulangu S, Dodd LE, Davey RT Jr, Tshiani Mbaya O, Proschan M, Mukadi D, Lusakibanza Manzo M, Nzolo D, Tshomba Oloma A, Ibanda A, Ali R, Coulibaly S, Levine AC, Grais R, Diaz J, Lane HC, Muyembe-Tamfum JJ; PALM Writing Group; Sivahera B, Camara M, Kojan R, Walker R, Dighero-Kemp B, Cao H, Mukumbayi P, Mbala-Kingebeni P, Ahuka S, Albert S, Bonnett T, Crozier I, Duvenhage M, Proffitt C, Teitelbaum M, Moench T, Aboulhab J, Barrett K, Cahill K, Cone K, Eckes R, Hensley L, Herpin B, Higgs E, Ledgerwood J, Pierson J, Smolskis M, Sow Y, Tierney J, Sivapalasingam S, Holman W, Gettinger N, Vallee D, Nordwall J; PALM Consortium Study Team. A Randomized, Controlled Trial of Ebola Virus Disease Therapeutics. N Engl J Med. 2019 Dec 12;381(24):2293-2303. doi: 10.1056/NEJMoa1910993. Epub 2019 Nov 27. PMID 31774950
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0003.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 681 patients enrolled, one pt was excluded due to a false + PCR result, 50 patients were enrolled prior to addition of the REGN-EB3 arm, and 7 patients underwent randomization during a 2-week period when ZMapp was unavailable. This led to 631 evaluable patients whose timing of enrollment permitted contemporaneous randomization to one of the three study arms versus the control (ZMapp) arm, as stipulated in version 3.0 of the protocol and at outlined in the Statistical Analysis Plan.
Pre-assignment Details: Statistical comparisons for efficacy between the three treatment arms and ZMapp as the control arm were limited to those time periods when contemporaneous enrollments could occur. So, for example, comparison between REGN-EB3 recipients and ZMapp recipients were limited to the time period beginning in January 2019 because that is when the REGN-EB3 arm was added as a fourth arm to the study.
Groups:
- Arm A: Remdesivir Plus Optimized Standard of Care (oSOC): Remdesivir: Administered intravenously with a loading dose on Day 1 (200 mg for adults and pediatric patients with body weight >= 40 kg and for pediatric patients weighing < 40 kg one loading dose of remdesivir 5 mg/kg) followed by 9 to 13 days of once-daily maintenance dosing starting on Day 2 and extending through Day 10 to 14 (100 mg for adults and pediatric patients with body weight >= 40 kg and for pediatric patients weighing < 40 kg remdesivir 2.5 mg/kg)
- Arm B: MAb114 Plus Optimized Standard of Care (oSOC): MAb114: 50 mg/kg of body weight administered intravenously on Day 1 as a single infusion
- Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC): REGN-EB3: 150 mg/kg of body weight administered intravenously on Day 1 as a single infusion
- Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC): ZMapp: Three doses of 50 mg/kg of body weight administered intravenously every third day beginning on Day 1
Period: Overall Study
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC)
Started | 177 | 176 | 158 (The REGN-EB3 arm was added in 1/2019 after the trial had initially begun in November 2018.) | 169
Completed | 169 (in 8/2019 the DSMB recommended further randomization only occur to the MAb114 and REGN-EB3 arms.) | 169 (in 8/2019 the DSMB recommended further randomization only occur to the MAb114 and REGN-EB3 arms.) | 154 (in 8/2019 the DSMB recommended further randomization only occur to the MAb114 and REGN-EB3 arms.) | 169 (in 8/2019 the DSMB recommended further randomization only occur to the MAb114 and REGN-EB3 arms.)
Not Completed | 8 | 7 | 4 | 0
Not completed — "not completed" simply refers to pts who could not be contemporaneously compared to the ZMapp arm | 8 | 7 | 4 | 0

BASELINE CHARACTERISTICS:
Population: as per the Statistical Analysis Plan, efficacy comparisons between each of the three investigational treatments and the ZMapp control arm were restricted to patients for whom contemporaneous randomization to the study arms was possible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC) | Total
Number analyzed (Participants) | 175 | 174 | 155 | 169 | 673
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (17.2) | 27.4 (18.5) | 28.2 (18.2) | 29.7 (16.8) | 28.8 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 98 | 91 | 87 | 374
  Male | 77 | 76 | 64 | 82 | 299
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 175 | 174 | 155 | 169 | 673
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Congo, The Democratic Republic of the | 175 | 174 | 155 | 169 | 673

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of Participants with Mortality by Day 28
Time Frame: 28 days
Population: patients randomized to receive one of the 4 investigational treatments
Measure: Number; unit: deaths
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC)
Number analyzed (Participants) | 175 | 174 | 155 | 169
deaths | 93 | 61 | 52 | 84

2. Secondary Outcome: Time in Days to First Negative Ebola Virus RT-PCR in Blood.
Description: This was a measure of the median number of days that it took for the serum PCR to first turn negative after having been positive throughout the patient's earlier course.
Time Frame: up to Day 28
Population: patients in all treatment arms who were randomized contemporaneously with those randomized to the control arm (Arm D).
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC)
Number analyzed (Participants) | 175 | 174 | 155 | 169
Days | NA [0 to 28] — Among patients in the remdesivir group, the estimated median time was actually more than 28 days because mortality exceeded 50% and expired patients were assigned a time of ">28 days". | 16 [0 to 28] | 15 [0 to 28] | 27 [0 to 28]

3. Secondary Outcome: Viremia as Determined by CTnp Values on PCR
Description: These are the median CTnp pCR values measured serially on the 4 treatment arms as per protocol.
  caveats: Undetectable ctNP values are imputed as ctNP=45.0 (the limit of detection). Missing values (due to gaps in sample collection, discharge, or death) are handled by carrying forward the last observation.
  The Day 28 visit includes a ±7-day visit window. The priority for defining the ctNP value for this timepoint, according to days post-randomization, is: 28, 27, 29, 26, 30, 25, 31, 24, 32, 23, 33, 22, 34, 21. For example, the ctNP result from the sample collected 26 days post-randomization will only be used for this timepoint if there are no sample results for 28, 27, or 29 days post-randomization.
Time Frame: Days 1, 2, 3, 4, 6, 8, 10, 14, and 28.
Population: these are the median CTnp PCR measurements performed serially on patients at defined timepoints on the 4 treatment arms
Measure: Median (Full Range); unit: median CTnp PCR values
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC)
Number analyzed (Participants) | 175 | 174 | 155 | 169
median CTnp PCR values
  ar randomization | 23.1 [10 to 45] | 23.4 [10 to 45] | 22.8 [10 to 45] | 23.1 [10 to 45]
  Day 1 | 22.2 [10 to 45] | 23.7 [10 to 45] | 23.3 [10 to 45] | 22.8 [10 to 45]
  Day 2 | 23.0 [10 to 45] | 25.1 [10 to 45] | 25.2 [10 to 45] | 23.7 [10 to 45]
  Day 3 | 23.7 [10 to 45] | 28.6 [10 to 45] | 28.1 [10 to 45] | 24.2 [10 to 45]
  Day 4 | 25.4 [10 to 45] | 30.9 [10 to 45] | 30.5 [10 to 45] | 25.7 [10 to 45]
  Day 6 | 28.6 [10 to 45] | 32.7 [10 to 45] | 32.7 [10 to 45] | 29.4 [10 to 45]
  Day 8 | 30.1 [10 to 45] | 34.4 [10 to 45] | 34.5 [10 to 45] | 32.2 [10 to 45]
  Day 10 | 31.6 [10 to 45] | 36.3 [10 to 45] | 36.3 [10 to 45] | 33.2 [10 to 45]
  Day 14 | 33.2 [10 to 45] | 39.1 [10 to 45] | 39.8 [10 to 45] | 35.2 [10 to 45]
  Day 28 | 37.6 [10 to 45] | 45.0 [10 to 45] | 45.0 [10 to 45] | 38.4 [10 to 45]

4. Secondary Outcome: Incidence of Serious Adverse Events/AEs
Description: The number of Serious Adverse Events that were tentatively ascribed to one of the four treatment arms by the site investigator and, upon extensive further review and adjudication by an independent Pharmacovigilance committee, were still felt potentially attributable to study drug as opposed to the underlying Ebola infection.
Time Frame: up to Day 58
Population: This table shows the number of SAEs adjudicated to be potentially related to study drug infusion for each of the four study arms. There were 4 SAEs reported in a total of 3 patients.
Measure: Number; unit: number of SAEs
Units Other Than Participants: doses
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC)
Number analyzed (Participants) | 175 | 174 | 155 | 169
Number analyzed (doses) | 1409 | 171 | 150 | 361
number of SAEs | 1 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: Patients were evaluated from time of randomization (Day 1) through Day 58 of study.
Description: Only SAEs that were felt by site investigators to be possibly study treatment-related and not due to underlying Ebola virus disease were reported, then subjected to rigorous review, additional data collection as necessary, and adjudication by an independent Pharmacovigilance team in order to separate those SAEs still most likely due to underlying Ebola infection from those potentially attributable to infusion(s) of one of the four assigned study drugs.
Arm/Group | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC)
All-Cause Mortality (participants affected / at risk) | 93/175 | 61/174 | 52/155 | 84/169
Serious Adverse Events (participants affected / at risk) | 1/175 | 0/174 | 0/155 | 2/169
Other Adverse Events (participants affected / at risk) | 6/175 | 1/174 | 2/155 | 6/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) (N=175) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) (N=174) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) (N=155) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC) (N=169)
death (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) — 4 events leading to death: in 1 patient it was worsening of GI symptoms reported as 2 separate events; in a second pt it was peri-infusional hypotension and hypoxia; in a third patient it was hypotension followed by cardiac arrest.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Remdesivir Plus Optimized Standard of Care (oSOC) (N=175) | Arm B: MAb114 Plus Optimized Standard of Care (oSOC) (N=174) | Arm C: REGN-EB3 Plus Optimized Standard of Care (oSOC) (N=155) | Control Arm (D): ZMapp Plus Optimized Standard of Care (oSOC) (N=169)
incomplete study drug infusion(s) (Surgical and medical procedures) | 6 (6) | 1 (1) | 2 (2) | 6 (6) — These are the number of investigational study drug infusions that were attempted but could not be completed due to various reasons.

LIMITATIONS AND CAVEATS:
By design, efficacy comparisons between the 3 investigational treatment arms and the ZMapp control arm were always restricted to those time periods when both ZMapp and the study drug were available, and there were brief periods when ZMapp became unavailable, accounting for why the total numbers compared between the arms are sometimes lower than the total number of enrolled patients. Also, the REGN-EB3 arm started enrolling later than the other three arms due to a protocol modification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03719586/Prot_SAP_ICF_000.pdf